CLINICAL TRIAL: NCT01024101
Title: Early Phase II Study of Weekly Paclitaxel (BMS-181339) in Patient With Advanced or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-372
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, IV, 100 mg/m², Weekly for 6 of 7 weeks, until disease progression or unacceptable toxicity became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of paclitaxel given weekly in patients with advanced or recurrent head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced head and neck cancer pretreated with surgery and/or radiotherapy and not suitable for further radical local treatment or patients with distant metastases who may have received no or one chemotherapy regimen

Exclusion Criteria:

* Patients with serious, uncontrolled medical illness

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Response rate [defined as total number of patients with complete and partial response divided by number of response-evaluable patients] based on predetermined evaluation criteria | Each 49 day course of treatment until withdrawal or unacceptable toxicity
Safety: incidence and severity of adverse events, laboratory test abnormalities | Each 49 day course of treatment until withdrawal or unacceptable toxicity

SECONDARY OUTCOMES:
Duration of response, defined as either Complete or Partial Response, based on Evaluation Criteria on Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer | Each 49 day course of treatment until withdrawal or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx